CLINICAL TRIAL: NCT05784688
Title: A Phase 1b/2a Study to Assess the Safety, Pharmacokinetics, and Preliminary Efficacy of TU2218, an Oral TGFβR Serine/Threonine Kinase Inhibitor, Administered in Combination With Pembrolizumab in Patients With Advanced Solid Tumors
Brief Title: Study of TU2218 in Combination With KEYTRUDA®(Pembrolizumab) in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: TiumBio Co., Ltd. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TUC1PI-02; MK-3475-E34 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2023-02-20; First posted 2023-03-27 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-02

CONDITIONS: Solid Tumor; Biliary Tract Cancer; Head and Neck Squamous Cell Carcinoma; Colorectal Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms; Squamous Cell Carcinoma of Head and Neck; Colorectal Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1b: TU2218 + KEYTRUDA® (Pembrolizumab) in solid tumor (Experimental): TU2218 orally and KEYTRUDA® (Pembrolizumab) intravenously administered daily for two weeks followed by one week to determine RP2DC.
  Interventions: Drug: TU2218 + KEYTRUDA® (Pembrolizumab)
- Phase 2a: TU2218 + KEYTRUDA® (Pembrolizumab) in Biliary Tract Cancer (BTC) (Experimental): TU2218 + KEYTRUDA® (Pembrolizumab) administered, orally BID, for 2 weeks followed by 1 week of rest in 3-week cycles for TU2218 and intravenous 200mg once every 3 weeks for KEYTRUDA® (Pembrolizumab)
  Interventions: Drug: TU2218 + KEYTRUDA® (Pembrolizumab)
- Phase 2a: TU2218 + KEYTRUDA® (Pembrolizumab) in Head and Neck Squamous Cell Carcinoma (HNSCC) (Experimental): TU2218 + KEYTRUDA® (Pembrolizumab) administered, orally BID, for 2 weeks followed by 1 week of rest in 3-week cycles for TU2218 and intravenous 200mg once every 3 weeks for KEYTRUDA® (Pembrolizumab)
  Interventions: Drug: TU2218 + KEYTRUDA® (Pembrolizumab)
- Phase 2a: TU2218 + KEYTRUDA® (Pembrolizumab) in ColoRectal Cancer (CRC) (Experimental): TU2218 + KEYTRUDA® (Pembrolizumab) administered, orally BID, for 2 weeks followed by 1 week of rest in 3-week cycles for TU2218 and intravenous 200mg once every 3 weeks for KEYTRUDA® (Pembrolizumab)
  Interventions: Drug: TU2218 + KEYTRUDA® (Pembrolizumab)

INTERVENTIONS:
Drug: TU2218 + KEYTRUDA® (Pembrolizumab) — TU2218: Orally administered KEYTRUDA® (Pembrolizumab): Intravenously administered

SUMMARY:
This study consists of phase 1b and 2a to evaluate safety, Pharmacokinetics, and efficacy of TU2218 in combination with Pembrolizumab in patients with advanced solid tumors.

DETAILED DESCRIPTION:
The primary objective of phase 1b is to determine the recommended phase 2 dose of the combination (RP2DC) of TU2218 given with pembrolizumab in advanced solid tumors.

The primary objective of phase 2a is to evaluate the efficacy of TU2218 administered in combination with pembrolizumab in selected advanced tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Male and females ≥18 years of age
2. Life expectancy ≥12 weeks as judged by the Investigator
3. Measurable disease as defined by RECIST v1.1
4. ECOG 0 or 1
5. Able to swallow capsules
6. For Phase 1b and 2a: histologically or cytologically documented advanced unresectable solid tumor for which no effective standard therapy exists, or that has progressed on or not tolerated prior standard therapy. If previously treated with an anti-PD-1/L1 mAb administered either as monotherapy, or in combination with other checkpoint inhibitors or other therapies, PD-1 treatment progression is defined by meeting all of the following criteria:

   1. Has received at least 2 doses of an approved anti-PD-1/L1 mAb
   2. Has demonstrated clinical progression after anti-PD-1/L1 mAb therapy
   3. Progressive disease has been documented within 16 weeks from the last dose of anti-PD-1/L1 mAb
7. For HNSCC cohort in Phase 2a: anti-PD-(L)1 agent-naïve metastatic or with unresectable, recurrent head and neck squamous cell carcinoma (HNSCC) whose tumors express programmed death ligand 1 (PD - L1) [combined positive score (CPS) ≥1] as determined by an FDA-approved test Or recurrent or metastatic head and neck squamous cell carcinoma (HNSCC) with disease progression on or after platinum-containing chemotherapy (as applicable).
8. For BTC cohort in Phase 2a: biliary tract cancer that has been locally advanced unresectable or metastatic or not tolerated prior standard first line chemotherapy and second line targeted therapy (as applicable).
9. For CRC cohort in Phase 2a: anti-PD-(L)1 agent-naïve colorectal adenocarcinoma of Proficient Mismatch Repair (pMMR)/Microsatellite Stable (MSS) subtype, as determined by an FDA-approved test, that has progressed on or not tolerated at least 2 lines of prior standard chemotherapy with biological agents where applicable. Patients with liver metastasis from primary CRC, as confirmed by RESIST v1.1, will be excluded from Phase 2a CRC cohort.
10. Adequate hematological function and coagulation defined by

    * ANC ≥1,500 cells/μL
    * Platelet count ≥100,000/μL
    * Hemoglobin ≥9.0 g/dL (criteria must be met without packed red blood cell transfusion within the prior 2 weeks. Participants can be on stable dose of erythropoietin [≥ approximately 3 months])
    * International normalized ratio ≤1.5 upper limit of normal (ULN)
11. Adequate hepatic and renal function

    * Total bilirubin ≤1.5 × ULN
    * AST and alanine aminotransferase (ALT) ≤2.5 × ULN; if liver metastases are present, then ≤5 × ULN is allowed.
    * Estimated creatinine clearance ≥60 mL/minute according to the Cockcroft Gault formula.
12. Able to understand and to comply with all protocol requirements, instructions, and restrictions. For Phase 2a, willing and able to provide archival tumor samples or undergo biopsy for biomarker testing during screening.
13. QTcF interval ≤470 msec on screening ECG.
14. Normal ejection fraction (within the reference range of the institution).
15. No concomitant anti-cancer treatments, including experimental agents for 5 half-lives for non-biological agents and a minimum of 4 weeks for any biologics prior to the start of treatment.
16. Resolution of any toxicity to maximum Grade 1 (except alopecia and Grade ≤2 neuropathy) prior to the start of treatment. Participants with endocrine-related AEs Grade ≤2 requiring treatment or hormone replacement are eligible.
17. Completion of radiotherapy (palliative or curative) at least 14 days prior to the start of treatment with resolution of any toxicity to maximum Grade 1. Participants must have recovered from all radiation-related toxicities and not require corticosteroids.
18. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

    1. Not a woman of childbearing potential (WOCBP) defined as all female after puberty unless they are postmenopausal for at least 1 year or are surgically sterile (hysterectomy or bilateral oophorectomy or tubal ligation).
    2. A WOCBP who has a negative serum pregnancy test within 3 days of the first administration of study treatment and agrees to follow contraceptive guidance during the treatment period and for at least 30 days after the last dose of TU2218 or until at least 120 days after the last administration of pembrolizumab, whichever comes later.

Exclusion Criteria:

1. Myocardial infarction within 6 months prior to screening, or pericardial effusion
2. History of cardiac or aortic surgery within 12 months
3. Unstable angina pectoris, cerebrovascular accident, transient ischemic attack, or symptomatic pulmonary embolism; deep venous thrombosis; arterial occlusive disease in the past 12 months
4. Congestive heart failure of New York Heart Association class III/IV
5. Major arrhythmia or abnormalities identified by ECG per Investigator's judgement
6. Uncontrolled hypertension (as defined by systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg) during the Screening Period.
7. Elevated Troponin I levels (Grade 3) at screening
8. Metastatic disease to the brain or central nervous system, carcinomatous meningitis, massive uncontrolled effusions (pleural, pericardial, peritoneal), and pulmonary lymphangitis
9. Known history of difficulty swallowing, malabsorption or other conditions that may reduce absorption of TU2218
10. Tumor that compresses or invades major blood vessels or tumor cavitation that in the opinion of the Investigator is likely to bleed
11. History of severe bleeding. Unable to stop anticoagulation therapy with heparin, low molecular weight heparin, vitamin K antagonists, anti-platelet agents, or factor Xa inhibitors throughout the study and for at least 28 days post the last dose of study treatment
12. Moderate or severe heart valve function defect including moderate or severe valve stenosis or regurgitation
13. Evidence or history of septal aneurysm, other heart aneurysm, or any aneurysm of the major vessels
14. Female participants must not be pregnant or at risk of becoming pregnant during the study. Fertile male and female participants must agree to use a highly effective method of birth control to avoid pregnancy (for female participants a double-barrier method of contraception, for male participants a condom with spermicide) or total abstinence from the time of providing informed consent until at least 30 days after the last dose of TU2218 or until at least 120 days after the last administration of Pembrolizumab, whichever comes later.
15. Female participants who are breastfeeding
16. For Phase 1b and BTC cohort in Phase 2a: discontinued prior therapy with an anti-PD-1, anti-PD-L1, or anti PD-L2 agent or with an agent directed to another stimulatory or co inhibitory T-cell receptor (e.g., CTLA-4, OX-40, CD137), due to an irAE.
17. For CRC and HNSCC cohorts in Phase 2a: received prior therapy with an anti-PD-1, anti PD-L1, or anti PD-L2 agent or an agent directed to another stimulatory or co inhibitory T-cell receptor (e.g., CTLA-4, OX-40, CD137).
18. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks (could consider shorter interval for kinase inhibitors or other short half-life drugs) prior to treatment.

    Note: Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy are eligible. Participants with endocrine-related AEs Grade ≤2 requiring treatment or hormone replacement are eligible.

    Note: If the participant had major surgery, the participant must have recovered adequately from the procedure and/or any complications from the surgery prior to starting study intervention.
19. Has received prior radiotherapy within 2 weeks of start of study treatment or have had a history of radiation pneumonitis.

    Note: Participants must have recovered from all radiation-related toxicities and not require corticosteroids. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-central nervous system (CNS) disease.
20. Has received or planned to receive any live or live-attenuated vaccine (e.g., measles, mumps, rubella or chickenpox) within 30 days prior to the first drug administration and while participating the study.

    Note: Administration of killed vaccines are allowed. Receipt of mRNA vaccine, including Coronavirus disease-2019 (COVID-19) vaccine, within 7 days prior to drug administration on Day 1 and during the first 2 cycles of study treatment will not be allowed
21. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent
22. Has had an allogeneic tissue/solid organ transplant
23. Received prior treatment targeting the signaling pathway of TGF-Beta
24. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study treatment
25. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ, excluding carcinoma in situ of bladder, that have undergone potentially curative therapy are not excluded
26. Has severe hypersensitivity (Grade ≥3) to Pembrolizumab and/or any of its excipients
27. Has an active autoimmune disease or history of autoimmune disease, except vitiligo, hypothyroidism or resolved childhood asthma/atopy, that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed
28. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
29. Has an active infection requiring systemic antibiotic therapy
30. Active and clinically significant bacterial, fungal, or viral infection, including known history of hepatitis B virus (HBV), known hepatitis C virus (HCV), known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome-related illness.

    Note: No testing for HBV, HCV, and HIV is required unless mandated by local healthy authority
31. Unable or unwilling to stop use of strong inhibitors of cytochrome P450 (CYP)1A2, 2C8 and 3A4, and strong inhibitors of P-gP and breast cancer resistance protein (BCRP) at least 8 days prior to and during study treatment in all Phase 1b dose escalation cohorts
32. Unable or unwilling to stop use of gastric pH elevating agents including proton pump inhibitors, H2-receptor antagonists and antacids at least 8 days prior to and during study treatment in all Phase 1b dose escalation cohorts
33. Has a history or current evident of any condition, therapy, or laboratory abnormality, or other circumstance that might confound the results of the study or interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating Investigator
34. Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study
35. Known history, or suspected hypersensitivity to any excipients of the clinical study treatments
36. Any other serious medical condition which in the Investigator's opinion would preclude safe participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Phase 1b: To determine the Recommended Phase 2 Dose of the Combination (RP2DC) of TU2218 given with Pembrolizumab in selected advanced solid tumors | During the first 21-day period (Cycle 1)
  At least 1 Dose limiting toxicity (DLT) during Cycle1
Phase 2a: To evaluate the efficacy of TU2218 by evaluating the Overall Response rate (ORR) of TU2218 administered in combination with Pembrolizumab in selected advanced solid tumors | 24 weeks
  ORR is defined as the proportion of patients with a best overall response of Complete response (CR) or Partial response (PR) according to RECIST v1.1 Efficacy analyses will be performed on both PP and ITT Efficacy Analysis Sets.

SECONDARY OUTCOMES:
Phase 1b and 2a: To further evaluate the safety and tolerability of TU2218 administered in combination with pembrolizumab. | approximately 13 months
  Incidence and severity of TEAEs, Incidence of Serious Adverse Events (SAE), Treatment Related Adverse Events (TRAE), and Adverse Events of Special Interest (AESI).
Phase 1b and 2a: The PK of TU2218 administered in combination with pembrolizumab | Cycle 1 (each cycle is 21 days)
  TU2218 plasma concentration
Time to Progression (TTP) | over 24 weeks
  TTP is defined as the time from first dose of study treatment to the date of first documented PD.
Duration of Response (DoR) | over 24 weeks
  DoR is defined as the duration between first documentation of CR or PR to first documentation of PD or death.
Disease Control Rate (DCR) | over 24 weeks
  DCR is defined as the proportion of participants with a best overall response of CR or PR or stable disease (SD)
Clinical Benefit Rate (CBR) | over 24 weeks
  CBR is defined as the proportion of participants with response or stabilization
Overall Survival (OS) | OS rate at 6 months = up to 24 weeks
  OS time is defined as the time from the date of first dose of study treatment to the date of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: TU2218, Study Director — TiumBio Co., Ltd.
Locations (11):
- United States (3):
  - NEXT Oncology, San Antonio, Texas
  - Hope Cancer Center, Tyler, Texas
  - Medical Oncology, Spokane, Washington
- South Korea (8):
  - CHA University Bundang Medical Center, Seongnam
  - Seoul National University Bundang Hospital, Seongnam
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - The Catholic University of Korea Seoul St. Mary Hospital, Seoul
  - The Catholic University of Korea St. Vincent's Hospital, Suwon

IPD SHARING:
Plan to Share IPD: No
We will make our final decision after EOP2 meeting.